CLINICAL TRIAL: NCT00765531
Title: Stone Disease in Children and Their Families
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Linda A Baker, Professor of Urology, Director of Pediatric Urology Research, University of Texas Southwestern Medical Center
Other Study IDs: STU 062011-081
Record Dates: First submitted 2008-09-30; First posted 2008-10-03 (Estimated); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Hypercalciuria; Urolithiasis
Keywords: Determine prevalence of genetic mutations in a population.; Identify stone formers w/significant family history.; follow a cohort of pediatric stone formers & their families.; Report long-term recurrence rates & therapeutic outcomes.
MeSH Terms: conditions — Hypercalciuria; Urolithiasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Testing group 1 - Patients with hypercalciuria and their families: 7 day diet and 44hr inpatient testing
- Testing group 2 - Patients with or without hypercalciuria and their families: 7 day diet and outpatient testing

SUMMARY:
The hypothesis of this study proposal is that pediatric urinary stone formers have genetic risk factors which predispose their urinary stone production. 50-60% of pediatric stone patients have a positive family history of urinary stone disease. Several genetic mutations have been identified which predispose patients to various types of urinary stones. These genetic mutations can also lead to other significant sequela besides stones, including osteopenia/osteoporosis (bone loss). Furthermore, metabolic abnormalities can be identified in more than 50% of pediatric stone formers, some of which can be improved and/or alleviated with medical intervention to help decrease rate of stone formation and the need for hospitalization and surgical intervention.

DETAILED DESCRIPTION:
Although more frequent in adults, urolithiasis (urinary stones) is not rare in children, accounting for an estimated 1 in 7,600 hospital admissions. Recent reports have demonstrated a rising incidence of urinary stones in children. The hypothesis of this study proposal is that pediatric urinary stone formers have genetic risk factors which predispose their urinary stone production. 50-60% of pediatric stone patients have a positive family history of urinary stone disease. Several genetic mutations have been identified which predispose patients to various types of urinary stones. These genetic mutations can also lead to other significant sequela besides stones, including osteopenia/osteoporosis (bone loss). Furthermore, metabolic abnormalities can be identified in more than 50% of pediatric stone formers, some of which can be improved and/or alleviated with medical intervention to help decrease rate of stone formation and the need for hospitalization and surgical intervention.

Independent of age, calcium is the main crystalline constituent of kidney stones in up to 80% of cases and calcium oxalate stones are the most common stone type. At all ages, hypercalciuria (urinary calcium excretion >4 mg/kg/d or urinary calcium / urinary creatinine > 0.2) is the most common metabolic cause of urolithiasis. Hypercalciuria is a common metabolic abnormality among patients who form calcium oxalate stones. Hypercalciuria can be primary (absorptive or renal) or secondary (resorptive). Primary absorptive hypercalciuria is the result of an increase in intestinal calcium absorption while primary renal hypercalciuria occurs when the kidneys leak calcium. Laboratory tests, including a serum parathyroid hormone level and urinary calcium excretion before and after dietary calcium restriction or load, are required to define which type of hypercalciuria is occurring. Secondary hypercalciuria may be the result of excessive sodium intake or induced by certain drugs. More commonly, secondary hypercalciuria is associated with other diseases (such as hypercalcemia, distal renal tubular acidosis, hyperparathyroidism, hypocitraturia, hypophosphatasia, Bartter's syndrome or prolonged immobilization). Whatever the cause, proper diagnosis and management of hypercalciuria in children is important since 50% may develop nephrocalcinosis and urolithiasis. In addition, vertebral bone loss has been reported in 30% of hypercalciuric children. In our patients who have undergone metabolic testing to date, approximately 50% have evidence of hypercalciuria.

Hypercalciuria resulting from increased absorption of calcium from the gut, termed absorptive hypercalciuria (AH), accounts for 45% of all reported cases of stone formation. AH has long been suspected to be genetic. More than 40% of first degree relatives of patients with hypercalciuria also have a history of urolithiasis. Over the last 10 years, investigators have sought to understand the molecular basis of this presumed genetic observation. The genotypes of individuals with hypercalciuria have been studied trying to associate polymorphisms in the vitamin D receptor gene with nephrolithiasis, but it seems vitamin D genotype has no clear influence on this phenotype. However, recently, a new candidate-gene was identified by Gitomer, et al which was linked to AH in Caucasian adults; it was mapped to chromosome 1q24. This gene has been putatively identified as a gut-specific soluble isoform of an adenylate cyclase which when mutated causes absorptive hypercalciuria. Four polymorphisms and two mutations have thus far been described; the presence of any of these 4 individual base substitutions yielded a 2.2 to 3.5-fold increase in estimated risk for absorptive hypercalciuria. These base changes were also associated with decreased spinal bone density and the occurrence of osteoporosis in the AH population. The incidence of gene mutations in this newly described AH gene has not been reported in children with either hypercalciuria, calcium oxalate stones or a positive family history.

In addition, novel candidate genes causing urolithiasis may be discovered during the duration of this study which would become subjects of investigation. Similarly, pedigrees from stone-forming probands affected in childhood have not been studied for medical outcomes, stone recurrence risks, or for novel gene searches. Unique pediatric stone cases that have been seen at Children's Medical Center include:

1. Xanthinuria (n=1)
2. Primary Hyperoxaluria, type 1 (n=1)
3. Cystinuria (n=3)
4. Hypocitraturia
5. Hyperoxaluria
6. Novel contiguous gene deletion syndrome with calcium nephrolithiasis (n=1)
7. Uric acid nephrolithiasis with metabolic syndrome (n=1)

Overall, although smaller numbers of affected patients are identified, the investigation of rare cases with a severe phenotype, which often first manifests in the pediatric population, may lead to a major disease discovery, as has been shown in many genetic diseases. Thus, we now broaden the scope of this research to include all pediatric stone-formers of all races and underlying metabolic and/or genetic abnormalities.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients of all races with a history of stone formation before age 20 years, patients with a history of stone formation between the ages of 4 and 19 years will be included regardless of current age or gender, healthy family members (>4 years of age to 75 years) of the probands will be invited to participate in the study and will be characterized as an affected or unaffected patient by the testing, and sex- and age-matched pediatric normal volunteers will also be recruited as controls.

Exclusion Criteria:

* Patients will be excluded with voiding dysfunction or metabolic disorders including renal tubular acidosis, chronic renal insufficiency, intestinal malabsorption (inflammatory bowel disease, history of ileal resection or bladder augmentation, and cystic fibrosis), hyperparathyroidism, prolonged immobilization, vitamin D excess, hypercalcemia, hypophosphatasia, Bartter's syndrome, high dose steroid therapy, prematurity, and chronic lasix use. Any child with a bleeding diathesis or who is immunocompromised will be excluded given the increased risks of drawing blood. Participants who have been on anti-seizure medication such as Topamax or other lithogenic drugs and anti-seizure medication will be excluded.

Ages: 4 Years to 20 Years | Sex: All
Age Groups: Child, Adult
Study Population: Individuals 4-20 years old of any sex with history of kidney stone formation and their family members.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Primary Completion 2022-09-26 (Actual); Study Completion 2022-12-05 (Actual)

PRIMARY OUTCOMES:
Urine calcium-creatinine ratio | 44 hours

CONTACTS AND LOCATIONS:
Overall Officials: Linda Baker, MD, Principal Investigator — Nationwide Children's Hospital

IPD SHARING:
Plan to Share IPD: No